CLINICAL TRIAL: NCT06358508
Title: Sapphire 3 - A Prospective, Open Label, Multi-center, Single Arm, Observational Study Designed to Evaluate the Acute Safety and Device Performance of the Sapphire 3 0.85-1.25 mm Coronary Dilatation Catheter in Predilatation of Chronic Total Occlusion (CTO) Lesions During Percutaneous Coronary Intervention.
Brief Title: Sapphire 3 CTO Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrbusNeich (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-0786
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases; Chronic Total Occlusion; Chronic Total Occlusion of Coronary Artery
Keywords: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases; Chronic Total Occlusion; Chronic Total Occlusion of Coronary Artery
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Sapphire 3 Coronary Dilatation Catheter (Experimental): Single arm with investigational Sapphire 3 Coronary Dilatation Catheters
  Interventions: Device: Sapphire 3 Coronary Dilatation Catheter

INTERVENTIONS:
Device: Sapphire 3 Coronary Dilatation Catheter — To pre-dilate Chronic Total Occlusion (CTO) lesions in coronary arteries during the subject's index procedure with Sapphire 3 0.85mm, 1.0mm, and 1.25mm diameter Coronary Dilatation Catheters.

SUMMARY:
A prospective, open label, multi-center, single arm, observational study designed to evaluate the acute safety and device performance of the Sapphire 3 0.85, 1.0 and 1.25mm diameter coronary dilatation catheter in predilatation of Chronic Total Occlusion (CTO) lesions during percutaneous coronary intervention.

One hundred seventy (170) subjects will be enrolled with a target of one hundred fifty-three (153) evaluable subjects by the angiographic core laboratory at up to 15 clinical sites with the Sapphire 3 0.85, 1.0 and 1.25mm diameter PTCA dilatation catheter to pre-dilate CTO lesions in coronary arteries during their index procedure. All subjects will be screened according to the protocol inclusion and exclusion criteria and will be followed through study completion, which is defined as 24-hours post-procedure or hospital discharge, whichever comes first.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedures.
3. Subject must agree not to participate in any other clinical study during hospitalization for the index procedure that would interfere with the endpoints of this study.
4. Subjects must have a single or double vessel coronary artery disease and clinical evidence of ischemic heart disease, such as stable / unstable angina or silent ischemia attributed to the CTO target vessel and is scheduled for clinically indicated percutaneous revascularization with planned stent placement during this index procedure.

   Angiographic Inclusion Criteria
5. Subject must have at least one de novo or restenotic lesion in native coronary arteries with Thrombolysis In Myocardial Infarction (TIMI) flow grade of 0 or 1 and is estimated to be at least 3 months in duration by clinical, angiographic, or electrocardiographic criteria.
6. A maximum of two lesions, including at least one target lesion, in up to two coronary arteries.
7. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion and must be deemed a clinical angiographic success by visual assessment.
8. The Target lesion is intended for stent placement during this index procedure.

Clinical Exclusion Criteria:

1. Subject with a known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, anti-platelet medications, or sensitivity to contrast media which cannot be adequately pre-medicated.
2. Evidence of acute myocardial infarction (MI) within 72 hours prior to the intended treatment defined as CK-MB or troponin greater than 1X the upper limit of normal (ULN).
3. Subject with known pregnancy or is nursing. Women of child- bearing potential should have a documented negative pregnancy test within 7 days before index procedure.
4. Planned or actual target lesion treatment prior to the use of the Study Device with an unapproved device, atherectomy, laser, cutting balloon or thrombectomy during the index procedure.
5. A serum creatinine level > 2.0 mg/dl within seven days prior to index procedure.
6. Cerebrovascular accident (CVA) within the past 6 months.
7. Active peptic ulcer or active gastrointestinal (GI) bleeding within the past 6 months.
8. Subject has a known left ventricular ejection fraction (LVEF) <30% (LVEF may be obtained at the time of the index procedure if the value is unknown, if necessary).

   Angiographic Exclusion Criteria
9. More than two lesions requiring treatment.
10. Unprotected left main coronary artery disease. (Greater than 50% diameter stenosis).
11. Coronary artery spasm of the target vessel in the absence of a significant stenosis.
12. Target lesion with angiographic presence of probable or definite thrombus of TIMI thrombus grade 3 or 4.
13. By visual estimation, target lesion involves a bifurcation requiring treatment with more than one stent or pre-dilatation of a side branch >2.25 mm in diameter.
14. Previous coronary interventional procedure of any kind within the 30 days prior to the procedure in the target vessel.
15. Target vessel with a patent bypass graft from prior coronary bypass surgery.
16. Previous stenting (drug-eluting or bare metal) in the target vessel unless all the following conditions are met:

    * It has been at least 9 months since the previous stenting.
    * That target lesion is at least 15 mm away from the previously placed stent. Total occlusions involving an in-stent segment are excluded.
    * The previously stented segment (stent plus 5 mm on either side) has no more than 40% diameter stenosis.
17. Non-target lesion to be treated during the index procedure meets any of the following criteria:

    * Located within a bypass graft (venous or arterial)
    * Left main location
    * Chronic total occlusion (CTO)
    * Is moderately to severely calcified.
    * Involves a bifurcation (e.g., bifurcations requiring treatment with more than 1 stent)
    * Treatment not deemed a clinical angiographic success

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Device Procedural Success | 24 hours post-procedure or hospital discharge, whichever comes first
  Device procedural success consisting of the following:
  * Successful delivery, inflation, deflation and withdrawal of the study balloon and after the guidewire has successfully crossed the CTO lesion into the true lumen of the vessel
  * No evidence of vessel perforation or dissections (Grade C or higher) related to the study balloon
  * Final TIMI flow grade of II or III at the conclusion of the PCI procedure

SECONDARY OUTCOMES:
Number of Participants With In-hospital Major Adverse Cardiac Events (MACE) | 24 hours post-procedure or hospital discharge, whichever comes first
  In-hospital Major Adverse Cardiac Events (MACE) which is a hierarchical composite of:
  * All death (cardiac and non-cardiac)
  * Myocardial infarction (MI)
  * Target Lesion Revascularization (TLR)
Number of Deaths (Cardiac and Non-Cardiac) | 24 hours post-procedure or hospital discharge, whichever comes first
  All death (cardiac and non-cardiac)
Number of Participants With Myocardial Infarctions (MI) | 24 hours post-procedure or hospital discharge, whichever comes first
  Myocardial Infarctions (MI)
Number of Participants With Target Lesion Revascularization (TLR) | 24 hours post-procedure or hospital discharge, whichever comes first
  Target Lesion Revascularization (TLR)
Number of Participants With In-hospital stent thrombosis (ST) Within the Target Vessel | 24 hours post-procedure or hospital discharge, whichever comes first
  In-hospital stent thrombosis (ST) Within the Target Vessel
Number of Participants With Clinically Significant Arrhythmias (Requiring Intervention) | 24 hours post-procedure or hospital discharge, whichever comes first
  Clinically Significant Arrhythmias (Requiring Intervention)
Number of Participants With Absence of Sapphire 3 Study Balloon Rupture | Peri-procedural
  Absence of Sapphire 3 Study Balloon Rupture
Number of Participants That Had Improvement in the Minimum Lumen Diameter (MLD) following use of Sapphire 3 catheter (independently measured by the Angiographic Core Lab using QCA) | Peri-procedural
  Improvement in Minimum Lumen Diameter (MLD) following use of Sapphire 3 catheter (measured by QCA).
  Improvement in MLD is defined as MLD post use of Sapphire 3 as greater than MLD from baseline.
Number of Participants With Technical Success | Peri-procedural
  Technical Success defined as Achievement of TIMI grade II or greater antegrade flow in all ≥2.5-mm distal branch(es) with <30% residual stenosis of the target CTO lesion at the completion of the procedure, (independently measured by the Angiographic Core Lab using QCA).

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute
Locations (14):
- United States (12):
  - Stanford Health Care, Stanford, California
  - Torrance Memorial Medical Center, Torrance, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - Atlanta VA Health Care System, Decatur, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital Heart and Vascular Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Washington, Seattle, Washington
- Spain (2):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Clinico Universitario de Valladolid, Valladolid